CLINICAL TRIAL: NCT03491228
Title: METRONIDAZOLE IV DRUG USE INVESTIGATION
Brief Title: Anaemetro I.V. Infusion 500mg Drug Use Investigation
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6831007
Record Dates: First submitted 2018-03-27; First posted 2018-04-09 (Actual); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Anaerobic Infection; Infectious Enterocolitis; Amebic Dysentery
MeSH Terms: conditions — Dysentery, Amebic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Secondary Data Collection Study; safety and effectiveness of Anaemetro under Japanese medical practice

ELIGIBILITY:
Inclusion Criteria:

* Patients who have not used metronidazole (injection) in the past, and have been given this drug for treatment of anaerobic infection, infectious enterocolitis, or amebic dysentery. Patients who have used metronidazole (oral agent and vaginal tablet) in the past are eligible, and should not be excluded from this study.

Exclusion Criteria:

* No exclusion criteria are set out in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who satisfy all of the inclusion criteria are subject to this study.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

RESULTS

PARTICIPANT FLOW:
Groups:
- ANAEMETRO Intravenous Infusion (Metronidazole): Participants who received ANAEMETRO Intravenous infusion as indicated in the approved local product document were observed for a period of maximum 8 weeks. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | ANAEMETRO Intravenous Infusion (Metronidazole)
Started | 107
Completed | 107
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 107 participants were enrolled in this study. There was no participant excluded from the baseline analysis.
Arm/Group | ANAEMETRO Intravenous Infusion (Metronidazole)
Number analyzed (Participants) | 107
Age, Customized [Number; unit: Participants]
  <15 years | 0
  ≥15 and <65 years | 40
  ≥65 years | 67
Sex/Gender, Customized [Number; unit: Participants]
  Male | 69
  Female | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Target Diseases [Number; unit: Participants] — Target diseases for this study were anaerobic infection, infectious enterocolitis, amebic dysentery, and the infection with both infectious enterocolitis and amebic dysentery.
  Participants
    Anaerobic infection | 74
    Infectious enterocolitis | 23
    Amebic dysentery | 7
    Infectious enterocolitis + amebic dysentery | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reaction (ADR)
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to ANAEMETRO Intravenous infusion in a participant who received ANAEMETRO Intravenous infusion. A serious ADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to ANAEMETRO Intravenous infusion was assessed by the physician.
Time Frame: Maximum 8 weeks
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received ANAEMETRO Intravenous infusion at least once.
Measure: Number; unit: Participants
Arm/Group | ANAEMETRO Intravenous Infusion (Metronidazole)
Number analyzed (Participants) | 107
Participants
  ADR | 7
  Serious ADR | 1

2. Secondary Outcome: Clinical Response Rate
Description: Clinical response of ANAEMETRO Intravenous infusion was evaluated comprehensively at the completion of the observation period, being assessed as "effective," "not effective," or "indeterminate" by the physician based on clinical symptoms.
  Clinical response rate, which was defined as the percentage of participants evaluated as "effective" over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI.
Time Frame: Maximum 8 weeks
Population: The clinical efficacy analysis set comprised of participants from the safety analysis set, excluding those with no information of clinical response or infections other than target disease. Participants evaluated as "indeterminate (n=12)" were excluded from the calculation.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ANAEMETRO Intravenous Infusion (Metronidazole)
Number analyzed (Participants) | 95
Percentage of Participants | 95.8 [89.6 to 98.8]

3. Secondary Outcome: Clinical Response Rates by Target Diseases
Description: Clinical response of ANAEMETRO Intravenous infusion was evaluated comprehensively at the completion of the observation period, being assessed as "effective," "not effective," or "indeterminate" by the physician based on clinical symptoms.
  Clinical response rate, which was defined as the percentage of participants evaluated as "effective" over the total number of assessable effectiveness analysis population, was presented along with the corresponding 2-sided 95% CI.
  Participants assessed as "effective" by the following target diseases were counted to assess whether they contribute to the clinical response: anaerobic infection, infectious enterocolitis, amebic dysentery, and the infection with both infectious enterocolitis and amebic dysentery.
Time Frame: Maximum 8 weeks
Population: The clinical efficacy analysis set comprised of participants from the safety analysis set, excluding those with no information of clinical response or infections other than target disease. Participants evaluated as "indeterminate (IND)" were excluded from the calculation.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | ANAEMETRO Intravenous Infusion (Metronidazole)
Number analyzed (Participants) | 95
Percentage of Participants
  Anaerobic infection (n=64)excluding IND(n=10): number analyzed (Participants) | 64
  Anaerobic infection (n=64)excluding IND(n=10) | 93.8 [84.8 to 98.3]
  Infectious enterocolitis (n=21) excluding IND(n=2): number analyzed (Participants) | 21
  Infectious enterocolitis (n=21) excluding IND(n=2) | 100.0 [83.9 to 100.0]
  Amebic dysentery (n=7): number analyzed (Participants) | 7
  Amebic dysentery (n=7) | 100.0 [59.0 to 100.0]
  Infectious enterocolitis + amebic dysentery (n=3): number analyzed (Participants) | 3
  Infectious enterocolitis + amebic dysentery (n=3) | 100.0 [29.2 to 100.0]

ADVERSE EVENTS:
Time Frame: Maximum 8 weeks
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both serious and non-serious events during the study.
Arm/Group | ANAEMETRO Intravenous Infusion (Metronidazole)
All-Cause Mortality (participants affected / at risk) | 3/107
Serious Adverse Events (participants affected / at risk) | 11/107
Other Adverse Events (participants affected / at risk) | 2/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ANAEMETRO Intravenous Infusion (Metronidazole) (N=107)
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 2
Multiple organ dysfunction syndrome (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ANAEMETRO Intravenous Infusion (Metronidazole) (N=107)
Nausea (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT03491228/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT03491228/SAP_001.pdf